CLINICAL TRIAL: NCT06936384
Title: The Investigation of the Effect of White Noise Sleep Mask on Patients' Sleep Quality and Comfort After Transurethral Resection of the Prostate (TUR-P) Surgery: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of White Noise Sleep Mask on Patients' Sleep Quality and Comfort After Transurethral Resection of the Prostate (TUR-P) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: White19999172490
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Surgical Procedures, Elective; Nurse Based Care Management
Keywords: White noise; sleep mask; surgical nursing; TUR-P; Transurethral Resection of the Prostate; surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In this group of patients, standard care will be applied during the postoperative period. Patients will sign an informed voluntary consent form before the surgery and fill out a patient information form.
  * Postoperative Day 1: Comfort level will be measured in the morning using the Richard Campbell Sleep Scale and the Visual Analog Scale (VAS). Patients will receive standard postoperative care without any additional interventions.
  * Postoperative Day 2: Reassessment will be done in the morning using the Richard Campbell Sleep Scale. Patients will be monitored according to standard care protocols during the postoperative process.
  * Postoperative Day 3: The final comfort assessment will be conducted using the Richard Campbell Sleep Scale and VAS.
  During this process, no additional mask or intervention will be applied; only routine postoperative care procedures will be followed.
- White Noise Sleep Mask Group (Experimental): White Noise Sleep Mask Group In this group, patients will be provided with a white noise sleep mask in accordance with the protocol determined for the postoperative period. Patients will sign an informed voluntary consent form before the surgery and fill out a patient information form.
  * Postoperative Day 1: Comfort level will be measured in the morning using the Richard Campbell Sleep Scale and the Visual Analog Scale (VAS). On the same day, in the morning, the nurse will recommend the patient use the white noise sleep mask twice a day for two hours. In the evening, the researcher will visit the hospital to ensure the mask is applied.
  * Postoperative Day 2: Reassessment will be done in the morning using the Richard Campbell Sleep Scale, and the mask usage will continue twice a day for two hours.
  * Postoperative Day 3: The final comfort assessment will be conducted using the Richard Campbell Sleep Scale and VAS.
  Interventions: Behavioral: In this group, patients will be provided with a white noise sleep mask in accordance with the protocol determined for the postoperative period. Patients will sign an informed voluntary consent form be

INTERVENTIONS:
Behavioral: In this group, patients will be provided with a white noise sleep mask in accordance with the protocol determined for the postoperative period. Patients will sign an informed voluntary consent form be — White Noise Sleep Mask Group In this group, patients will be provided with a white noise sleep mask in accordance with the protocol determined for the postoperative period. Patients will sign an informed voluntary consent form before the surgery and fill out a patient information form.
  Arms: White Noise Sleep Mask Group

SUMMARY:
One of the greatest challenges patients face in the postoperative period is the deterioration of sleep quality. Decreased sleep quality in the postoperative period is commonly observed due to pain, stress, anxiety, hospital environment noise, and environmental factors. Poor sleep quality can have negative effects on tissue healing, immune system activity, and overall well-being.

DETAILED DESCRIPTION:
Transurethral prostate resection (TUR-P) is one of the most commonly performed surgical procedures for the treatment of benign prostatic hyperplasia (BPH). Patients undergoing TUR-P surgery may experience sleep problems in the postoperative period due to the use of urinary catheters, discomfort in the pelvic region, frequent urination urges, bladder spasms, and factors related to the hospital environment. Improving comfort and sleep quality during the recovery process for these patients may contribute to the improvement of their overall health status. White noise is a type of sound that contains all frequencies at equal intensity and helps mask environmental noises, allowing individuals to have a more restful sleep experience . Literature has reported positive effects of white noise, such as increasing sleep duration, reducing sleep onset time, and decreasing nighttime awakenings. Studies have shown that the use of white noise, particularly in hospital settings, improves sleep quality. For example, a study conducted in an intensive care unit reported that white noise significantly improved sleep quality by masking disruptive sounds in the hospital environment. Similarly, findings suggest that the use of white noise in the postoperative period helps patients experience deeper and uninterrupted sleep. White noise sleep masks can support the sleep process by both blocking environmental sounds and minimizing visual stimuli. Considering that factors such as lighting and noise in the hospital environment can lead to sleep disturbances, it is believed that white noise sleep masks may be effective in improving sleep quality in the postoperative period. This study aims to evaluate the effect of using a white noise sleep mask on sleep quality and comfort in patients after TUR-P surgery. The current literature on non-pharmacological approaches to improving sleep quality in patients after TUR-P is limited. Therefore, evaluating the effectiveness of white noise sleep masks is an important new intervention area that may contribute to postoperative patient care

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* No hearing and perception problems,
* No visual impairment,
* Will undergo elective TUR-P

Exclusion Criteria:

* Use of any sleep/hypnotic medication or antidepressants before or after the procedure,
* Having a psychiatric disorder.
* Urgent surgery
* Suffering from sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-19 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale-Comfort | Postop day 1
  It is a form consisting of a 10 cm long horizontal line used to assess the subjective discomfort of patients. It is used to determine many conditions. VAS is a measurement tool that is 0-10 cm (0-100 mm) long. This measurement tool can be used horizontally or vertically. The scale starts with "I am not comfortable at all" and ends with "I am perfectly comfortable".
Visual Analog Scale-Comfort | Postop day 3
  It is a form consisting of a 10 cm long horizontal line used to assess the subjective discomfort of patients. It is used to determine many conditions. VAS is a measurement tool that is 0-10 cm (0-100 mm) long. This measurement tool can be used horizontally or vertically. The scale starts with "I am not comfortable at all" and ends with "I am perfectly comfortable".
Sleep Quality | Postop day 1
  The scale, which consists of 6 items in total, is evaluated on a chart with numbers between 0 and 100, each of the 6 items evaluating the depth of night sleep, the time to fall asleep, the frequency of waking up, the time to stay awake when waking up, the quality of sleep and the level of noise in the environment. Scores in the range "0-25" indicate very poor sleep and scores in the range "76-100" indicate very good sleep. The increase in the scores on the scale increases in direct proportion to the sleep quality of the participants.
Sleep Quality | Postop day 2
  The scale, which consists of 6 items in total, is evaluated on a chart with numbers between 0 and 100, each of the 6 items evaluating the depth of night sleep, the time to fall asleep, the frequency of waking up, the time to stay awake when waking up, the quality of sleep and the level of noise in the environment. Scores in the range "0-25" indicate very poor sleep and scores in the range "76-100" indicate very good sleep. The increase in the scores on the scale increases in direct proportion to the sleep quality of the participants.
Sleep Quality | Postop day 3
  The scale, which consists of 6 items in total, is evaluated on a chart with numbers between 0 and 100, each of the 6 items evaluating the depth of night sleep, the time to fall asleep, the frequency of waking up, the time to stay awake when waking up, the quality of sleep and the level of noise in the environment. Scores in the range "0-25" indicate very poor sleep and scores in the range "76-100" indicate very good sleep. The increase in the scores on the scale increases in direct proportion to the sleep quality of the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Cansu Yeniğün, Antalya, Kumluca, Turkey (Türkiye)